CLINICAL TRIAL: NCT04257435
Title: The Utility of Positive Psychology in Military TBI Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit individuals for the study
Sponsor: Fort Belvoir Community Hospital (U.S. Federal Agency)
Collaborators: The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The UPP Study; WRNMMC-2019-0216 (Other: WRNMMC)
Record Dates: First submitted 2019-03-18; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Behavioral Health Treatment (Active Comparator)
  Interventions: Behavioral: Traditional Behavioral Health Treatment
- Positive Psychological Group Treatment (Experimental)
  Interventions: Behavioral: Positive Psychological Group Treatment; Behavioral: Traditional Behavioral Health Treatment

INTERVENTIONS:
Behavioral: Positive Psychological Group Treatment — Positive psychological group treatment will involve engagement in traditional behavioral health treatment, as well as a group treatment focusing on previously researched exercises that have been demonstrated to relate to reduced depression and increased positive emotionality (Seligman, Rashid, Parks, et al., 2005; Seligman, Rashid, & Parks, 2006; Rashid, 2015).
  Arms: Positive Psychological Group Treatment
Behavioral: Traditional Behavioral Health Treatment — Treatment will include traditional individual behavioral health treatment, involving CBT-based therapeutic interventions for presenting diagnoses (typically depression, anxiety, or PTSD-related symptomatology).

SUMMARY:
Service members and veterans (SMVs) report more persisting symptoms following traumatic brain injury (TBI) compared to civilian populations (Ommaya, Ommaya, Dannenber, & Salazar, 1996). Therefore, it is important to utilize interventions that reduce psychological impairments and increase resiliency during military TBI rehabilitation. Unlike traditional behavioral health treatments that focus on reducing maladaptive behaviors and negative thoughts, positive psychological treatments focus on increasing positive emotions to increase well-being. There is substantial growing evidence demonstrating that cultivating positive emotions is preventative and improves resiliency and psychological (Bolier et al., 2013; Sin & Lyumbomirsky, 2009), cognitive (Estrada, Isen, & Young, 1997; Ashby & Isen, 1999; Isen & Daubman, 1984; Isen, Daubman, & Nowicki, 1987; Fredrickson & Branigan, 2001), and health outcomes (Pressman & Cohen, 2005). This study will examine the effectiveness of traditional behavioral health treatment versus behavioral health treatment with an added positive psychological group treatment in terms of psychological, cognitive, and health outcomes during TBI rehabilitation. The hypothesis is that SMV's with TBI will experience improved outcomes with added positive psychological treatment compared to traditional behavioral health treatment alone.

There will be about 100 people taking part in the study, randomly assigned to either a traditional behavioral health treatment group or an alternative behavioral health treatment group (therefore, up to 50 people will be enrolled in each) at the Fort Belvoir Intrepid Spirit Center over a period of 30 months. Study participants will be randomly assigned to groups, and over 3 months the study procedures include participating in group behavioral health treatment and/or individual behavioral health treatment and completing pre/post-treatment questionnaires focusing on psychological, cognitive, and health outcomes. The behavioral health intervention has not been well-studied; thus, the behavioral health intervention is considered experimental for the treatment of psychological symptoms. Additionally, the impact on other areas of functioning (i.e., cognitive functioning and overall health) is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Documented mild TBI or moderate TBI.
* Individual is recommended to have a Behavioral Health provider at ISC Fort Belvoir for general TBI-related psychological impairments.
* Individual has decision making capacity for informed consent based on medical provider clinical judgement and initial evaluation.
* Individual scored a 14 or lower on the Patient Health Questionnaire-9, indicating no worse than moderate depressive symptoms.
* Individual is 18 years or older.
* Individual is Defense Enrollment Eligibility Reporting System-eligible.

Exclusion Criteria:

* Individuals with severe depressive symptoms (PHQ-9 score above 14).
* Documented severe traumatic brain injury.
* Minors and pediatric populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in Positive Affect | Pre-treatment and at 3 month follow-up following study completion
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire on which participants rate adjectives of positive and negative feelings on a scale from 1 (very slightly/not at all) to 5 (extremely) according to how much they are currently experiencing that feeling. The sum of the positive items provides a measure of positive affect at each time point.

SECONDARY OUTCOMES:
Change in Hope | Pre-treatment and at 3 month follow-up following study completion
  The Hope Scale is a 12-item self-report questionnaire examining a patient's willful sense of determination to meet goals and a patient's perceived availability of ways to attain a goal. Higher ratings indicate greater hope at time of measurement.
Change in Life Satisfaction | Pre-treatment and at 3 month follow-up following study completion
  The General Life Satisfaction scale from NIH Toolbox is a 5-item scale designed to measure global cognitive judgments of one's life satisfaction. Participants indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. The total summed score will indicate satisfaction with life.
Change in Depression | Pre-treatment and at 3 month follow-up following study completion
  The Patient Health Questionnaire-9 is a 9-item measure given to screen for the presence and severity of depression. The total summed score indicates level of depression.
Change in Perceived Stress | Pre-treatment and at 3 month follow-up following study completion
  The Perceived Stress scale from NIH Toolbox is a 10-item measure given to assess perceptions about the nature of events and their relationship to the values and coping resources of an individual. Participants indicate how often behaviors and/or thoughts related to stress have occurred on a 5-point scale (Never to Very Often). The total summed score indicates overall perceived stress.
Change in Cognitive Functioning | Pre-treatment and at 3 month follow-up following study completion
  The Cognitive Functioning scale from Neuro QOL includes 8 items measuring perceived difficulties in cognitive abilities (e.g., memory, attention, and decision making, or in the application of such abilities to everyday tasks (e.g., planning, organizing, calculating, remembering and learning). Items are answered as 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=Very much. The total summed score indicates perceived cognitive functioning.
Change in Fatigue | Pre-treatment and at 3 month follow-up following study completion
  The Fatigue scale from Neuro QOL includes 8 items measuring sensations of tiredness to exhaustion that decreases one's capacity for physical, functional, social, and mental activities. Items are rated on a 5-point scale ranging from never to always. The total summed score indicates level of fatigue.
Change in Pain Intensity | Pre-treatment and at 3 month follow-up following study completion
  The Pain Intensity Survey from NIH Toolbox includes one item for self-reporting a participant's level of pain in the past seven days, ranging from 0 (no pain) to 10 (worst imaginable pain).
Change in Negative Affect | Pre-treatment and at 3 month follow-up following study completion
  The Positive and Negative Affect Schedule (PANAS) is a self-report questionnaire on which participants rate adjectives of positive and negative feelings on a scale from 1 (very slightly/not at all) to 5 (extremely) according to how much they are currently experiencing that feeling. The sum of the negative items provides a measure of negative affect at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Elion, PhD, Principal Investigator — Fort Belvoir Community Hospital
Locations (1):
- Fort Belvoir Community Hospital, Fort Belvoir, Virginia, United States

REFERENCES:
- [Background] Bolier L, Haverman M, Westerhof GJ, Riper H, Smit F, Bohlmeijer E. Positive psychology interventions: a meta-analysis of randomized controlled studies. BMC Public Health. 2013 Feb 8;13:119. doi: 10.1186/1471-2458-13-119. PMID 23390882
- [Background] Estrada C, Isen AM, & Young MJ (1997). Positive affect facilitates integration of information and decreases anchoring in reasoning among physicians. Organizational Behavior and Human Decision Processes, 72, 117-135.
- [Background] Ashby FG, Isen AM, Turken AU. A neuropsychological theory of positive affect and its influence on cognition. Psychol Rev. 1999 Jul;106(3):529-50. doi: 10.1037/0033-295x.106.3.529. PMID 10467897
- [Background] Isen, AM, & Daubman, KA (1984). The influence of affect on categorization. Journal of Personality and Social Psychology, 47(6), 1206-1217.
- [Background] Isen AM, Daubman KA, Nowicki GP. Positive affect facilitates creative problem solving. J Pers Soc Psychol. 1987 Jun;52(6):1122-31. doi: 10.1037//0022-3514.52.6.1122. PMID 3598858
- [Background] Fredrickson, BL, Branigan, A (2001). Positive emotions. In: Mayne, T.J.; Bonnano, G.A., editors. Emotion: Current issues and future developments. New York: Guilford Press, 123-151.
- [Background] Pressman SD, Cohen S. Does positive affect influence health? Psychol Bull. 2005 Nov;131(6):925-971. doi: 10.1037/0033-2909.131.6.925. PMID 16351329
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Seligman MEP, Rashid T, Parks AC. Positive psychotherapy. Am Psychol. 2006 Nov;61(8):774-788. doi: 10.1037/0003-066X.61.8.774. PMID 17115810
- [Background] Rashid, T (2015). Positive psychotherapy: A strength-based approach. The Journal of Positive Psychology, 10 (1), 25-40.